### КОМИТЕТ ПО БИОЭТИКЕ ПРИ САМАРСКОМ ГОСУДАРСТВЕННОМ МЕДИЦИНСКОМ УНИВЕРСИТЕТЕ

443079, г. Самара, ул. Гагарина, д.20

Тел. 8 (846) 374-10-04 (доб. 4200)

## ВЫПИСКА из ПРОТОКОЛА № 253

заседания Комитета по биоэтике при Самарском государственном медицинском университете от «14» сентября 2022 г.

Присутствовали члены Комитета по биоэтике: Волова Л.Т. - председатель, Антимонов А.В. – заместитель председателя, ответственный за клинические исследования, Ардашкин А.П., Кузнецов С.И., Шмелев И.А., Белоконев В.И., Санталова Г.В., Россинская В.В., Максименко Н.А., Резников В.Е. Кворум имеется.

Заседание состоялось 14.09.2022 г. в 12.00 ч. по адресу: ул. Гагарина, д.20.

#### СЛУШАЛИ:

Рассмотрение вопроса о соответствии этическим требованиям научного исследования аспиранта кафедры педиатрии ИПО СамГМУ Скворцовой О.В. «Клинико-метаболическая, иммунологическая и микробиологическая характеристика как основа дифференцированной тактики ведения детей с ожирением».

# На рассмотрение предоставляются следующие документы:

- 1. Протокол исследования.
- 2. Сведения о квалификации исследователя.
- 3. Сведения о квалификации научного руководителя.
- 4. Декларация о соблюдении международных и российских этических принципов и норм.
- 5. Индивидуальная регистрационная карта случая.
- 6. Информированное согласие пациента.

## ОГОВОРКА О КОМПЕТЕНТНОСТИ КОМИТЕТА

Предметом рассмотрения Комитета являются этические аспекты клинического исследования в соответствии с Этическим кодексом Российского врача, утвержденного на 4-й Конференции Ассоциации врачей России, Хельсинкской декларацией Всемирной медицинской ассоциации, п.15 ст. 37 ФЗ "Об основах охраны здоровья граждан в Российской Федерации" от 21.11.2011 № 323-ФЗ.

### постановили:

одобрить научное исследование Скворцовой О.В. «Клинико-метаболическая, иммунологическая и микробиологическая характеристика как основа дифференцированной тактики ведения детей с ожирением» как соответствующее этическим нормам.

Председатель Комитета по биоэтике, Д.м.н., профессор

Л.Т. Волова